CLINICAL TRIAL: NCT07174752
Title: Esthetic Evaluation of Non-Submerged De-Epithelialized Free Gingival Graft (Ns-dFGG) Versus Conventional Free Gingival Graft (cFGG) for the Augmentation of The Keratinized Mucosa: Randomized Controlled Clinical Trial
Brief Title: Non-Submerged De-Epithelialized Free Gingival Graft Versus Conventional Free Gingival Graft
Acronym: Ns-dFGG; cFGG
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: October University for Modern Sciences and Arts (Other)
Responsible Party: Principal Investigator, Dalia Khorshed, Masters candidate, October University for Modern Sciences and Arts
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 61124; Ethical committee (Other: 6 October university for Modern Sciences and Arts)
Record Dates: First submitted 2025-08-06; First posted 2025-09-16 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-08

CONDITIONS: Deficient Keratinized Mucosa

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ns-dFGG (Active Comparator): This arm will receive a Non-Submerged De-Epithelialized Free Gingival Graft for for the Augmentation of The Keratinized Mucosa
  Interventions: Procedure: Non-Submerged De-Epithelialized Free Gingival Graft
- FGG (Active Comparator): This arm will receive a Conventional Free Gingival Graft for for the Augmentation of The Keratinized Mucosa
  Interventions: Procedure: Conventional FGG

INTERVENTIONS:
Procedure: Non-Submerged De-Epithelialized Free Gingival Graft — The Free gingival graft will be de-epithelialized and fixed at the recipient site in a non-submerged manner to increase the keratinized mucosa
  Arms: Ns-dFGG
Procedure: Conventional FGG — The Free gingival graft will be fixed at the recipient site to increase the keratinized mucosa
  Arms: FGG

SUMMARY:
The goal of this (study type: RCT) is to learn if the use of the non-submerged de-epithelized FGG will result in better esthetic outcomes in adults. The main questions that it aims to answer are:

* Does this procedure increase the width of keratinized tissue?
* Does this procedure increase the depth of the vestibule? Researchers will compare this technique with the gold standard using the FGG to evaluate which technique provides better esthetics.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients: 18-60.
* Insufficient width of keratinized mucosa, that is less than 2 mm.
* Lower anterior areas.
* Good oral hygiene.

Exclusion Criteria:

* Systemic conditions that prevent the patient from undergoing minor oral surgical procedures or hinder the healing process.
* Patient undertaking radiotherapy or chemotherapy.
* Smokers.
* Pregnant females

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-12-29 (Actual); Primary Completion 2026-07-29 (Estimated); Study Completion 2026-12-29 (Estimated)

PRIMARY OUTCOMES:
Esthetic Evaluation of Non-Submerged De-Epithelialized Free Gingival Graft (Ns-dFGG) Versus Conventional Free Gingival Graft (cFGG) for the Augmentation of The Keratinized Mucosa | 6 months
  The professional esthetic evaluation will be done using the root coverage esthetic score (RES) by(Cairo et al.,2009).
  Standardized Clinical photographs will be taken at 6 months, where they will evaluate:
  Color matching: Score 0, & Score 1: Regarding the color matching to the normal gingiva Soft tissue texture: Score 0, & Score 1: If there is scar formation or keloid appearance Muco-gingival junction (MGJ) alignment: Score 0, & Score 1:If the MGJ is or isn't aligned that of the adjacent teeth
Esthetic Evaluation of Non-Submerged De-Epithelialized Free Gingival Graft (Ns-dFGG) Versus Conventional Free Gingival Graft (cFGG) for the Augmentation of The Keratinized Mucosa | 6 months
  The patient esthetic evaluation will evaluated at 6 months during the follow-up based on the Visual Analogue Scale(VAS). They will select among 100 scores of color matching: Score 0(Very bad) 50(Average) 100(Excellent)

CONTACTS AND LOCATIONS:
Locations (1):
- October University for modern sciences and arts (MSA University), Giza, Egypt

IPD SHARING:
Plan to Share IPD: No
collective data of the study groups will be available